CLINICAL TRIAL: NCT00803140
Title: A Pilot Study Comparing Cutaneous Scarring When Scalpel Versus Cautery is Used to Make Skin Incisions
Brief Title: Cutaneous Scarring of Scalpel Versus Cautery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual of subject enrollment.
Sponsor: Scott and White Hospital & Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81818CSSvC
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Scars
Keywords: scarring
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cautery Arm (Active Comparator): Cautery to make skin incision
  Interventions: Procedure: Cautery vs Active Control Arm (Scalpel)
- Scalpel Incision (Active Comparator): Scalpel to make skin incision
  Interventions: Procedure: Cautery vs Active Control Arm (Scalpel)

INTERVENTIONS:
Procedure: Cautery vs Active Control Arm (Scalpel) — Interventions: The cautery used will be the standard operating room monopolar cautery used at our institution. The cautery will be used on a "cut" setting of 20 with a blend setting of zero (pure cut). A standard protected needle tip cautery will be used.
  A #15 blade carbon steel scalpel blade will be used on ½ of the incision; a cautery device with the above-mentioned settings will be used on the other ½ of the wound. The patient will be randomly assigned to receive the cautery incision on the left or right side. The same surgeon will make all of the skin incisions and perform the skin closures in order to provide as much standardization as possible.
  The closure will be standardized.
  Other Names: bovie

SUMMARY:
Cutaneous scarring after elective surgery is a concern for surgeons of all types, perhaps even more so to plastic surgeons. Cautery is often used on the "cut" setting to make or extend incisions; however very few studies have looked at the results of these scars. The investigators' study aims are to compare standard scalpel incisions versus cautery incisions and to objectively compare the resultant scars in a prospective, randomized, controlled fashion.

DETAILED DESCRIPTION:
Rationale: Most surgeons at some point have used the "cut" setting on a cautery device to make or extend an incision. Anecdotally, there does not appear to be a noticeable difference in the scarring. This opinion, however is not shared by all surgeons.

Review of the literature reveals a paucity of evidence supporting the use of cutting cautery vs. standard, scalpel incision. A study that objectively, prospectively, and randomly compares the scars between these two methods has the potential to alter the doctrine of scalpel incisions, potentially saving money, and allowing a safer operating room environment (one free of scalpels in some cases).

Objectives: To objectively compare the cutaneous scars resulting from scalpel versus cutting cautery incisions using a subjective and objective scar measurement tool.

Methodology:

Research Design: This study will be a Blinded, Prospective, Randomized Controlled Trial.

Research Participants:

Comparison Information: The patient will have ½ of the incision performed with standard scalpel incision, and the contralateral ½ of the incision with cutting cautery incision. The sides will be randomized using a random number generator. For purposes of this study, the right side of the incision is defined as the patient's right side and the left side of the incision is defined as the patient's left side.

Criteria for Discontinuation: The study will be discontinued if it becomes obvious that the cautery ½ of the incision develops increased complications relating to infections, wound breakdown, or scarring.

Observations: The patients will follow up after surgery for evaluations at 2 weeks, 3 months, 6 months, and 12 months. Patients, physicians and a blinded independent observer will evaluate the scars using a visual analogue scale at 2 weeks, 3 months, 6 months and 12 months. Also, at 12 months, the Patient and Observer Scar Assessment Tool will be used to evaluate all scars in order to provide objective and subjective scar evaluation. The subject, surgeon and blinded observer will complete this evaluation.

Sample Size: 10 patients will be enrolled in our study. The data gathered from this pilot study should provide us with the data necessary to perform a power and sample size calculation for a future randomized controlled trial.

Date Management and Analysis: At postoperative follow up visits (2 weeks +/- 4 days, 3 months +/- 2 weeks, 6 months +/- 2 weeks), the patient, physician and independent observer will evaluate the scar subjectively using a visual analogue scale measuring 10 cm in length. One side of the scale (the side nearest 0) will imply the poorest scar imaginable; the opposite side will represent the best. Measurements will be taken regarding width, and observations regarding erythema and pigment will be noted.

At the 12 month postoperative follow up, the Patient and Observer Scar Assessment Tool will be used to compare the scars in order to provide both subjective and objective data.

Ethical Considerations

Protection of Human Subjects: Approval from the IRB will be obtained prior to beginning this study. All investigators have met federal and institutional educational requirements for Human Subjects Protection.

Patients will be offered scar revisions at no additional costs to the patient on the "test" side. These scar revisions will be offered at 1 year if necessary.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria:

1. Patients undergoing primary, elective panniculectomy.
2. Patients must voluntarily be enrolled in the study after informed consent.
3. Patients must be in relative good health and have adequate nutrition.
4. Patients of all races and genders will be included.
5. Patients must agree to refrain from the use of topical scar products during the study period.

Exclusion Criteria:

1. Under the age of 18 years old
2. Patients with previous history of hypertrophic or keloid scarring
3. Patients presenting for scar revision
4. Patients presenting for a non-elective surgery
5. Patients with chronic immunosuppression or wound healing problems
6. Currently taking medications that interfere with wound healing such as corticosteroids, anti-coagulants (aspirin or NSAIDs), vasoconstricting agents (adrenaline or ergotrate), anti-cancer drugs, or colchicine for gout,
7. Use of any tobacco products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the Vancouver Scar Scale | 12 months

SECONDARY OUTCOMES:
Visual scar scale done by both the subject and an independent observer | 2 week
Visual scar scale done by both the subject and an independent observer | 3 months
Visual scar scale done by both the subject and an independent observer | 6 months
Visual scar scale done by both the subject and an independent observer | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Raman C Mahabir, MD, Principal Investigator — Scott and White Hospital & Clinic
Locations (1):
- Scott and White Hospital and Clinic, Temple, Texas, United States

REFERENCES:
- [Background] Nguyen DQ, Potokar T, Price P. A review of current objective and subjective scar assessment tools. J Wound Care. 2008 Mar;17(3):101-2, 104-6. doi: 10.12968/jowc.2008.17.3.28666. PMID 18376650
- [Background] van Zuijlen PP, Angeles AP, Kreis RW, Bos KE, Middelkoop E. Scar assessment tools: implications for current research. Plast Reconstr Surg. 2002 Mar;109(3):1108-22. doi: 10.1097/00006534-200203000-00052. PMID 11884845
- [Background] Papay FA, Stein J, Luciano M, Zins JE. The microdissection cautery needle versus the cold scalpel in bicoronal incisions. J Craniofac Surg. 1998 Jul;9(4):344-7. doi: 10.1097/00001665-199807000-00010. PMID 9780929
- [Background] Sheikh B. Safety and efficacy of electrocautery scalpel utilization for skin opening in neurosurgery. Br J Neurosurg. 2004 Jun;18(3):268-72. doi: 10.1080/02688690410001732715. PMID 15327229
- [Background] Molgat YM, Pollack SV, Hurwitz JJ, Bunas SJ, Manning T, McCormack KM, Pinnell SR. Comparative study of wound healing in porcine skin with CO2 laser and other surgical modalities: preliminary findings. Int J Dermatol. 1995 Jan;34(1):42-7. doi: 10.1111/j.1365-4362.1995.tb04379.x. PMID 7896488
- [Background] Middleton WG, Tees DA, Ostrowski M. Comparative gross and histological effects of the CO2 laser, Nd-YAG laser, scalpel, Shaw scalpel and cutting cautery on skin in rats. J Otolaryngol. 1993 Jun;22(3):167-70. PMID 8371327